CLINICAL TRIAL: NCT00541710
Title: Genistein Use in Postmenopausal Women With Metabolic Syndrome
Brief Title: Effect of Genistein in Women With Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Messina (Other)
Collaborators: Ministry of Education, Universities and Research, Italy (Other)
Responsible Party: Principal Investigator, Rosario D'anna, Associate Professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RODA-12254; 20073XZSR3 (Other Grant/Funding Number: MIUR Italian Ministry of Research)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome
Keywords: menopause; genistein; pre-diabetes
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Placebo Comparator): Placebo tablets. All participants were counseled on an moderate hypocaloric, Mediterranean-style diet composed of 25% to 30% energy from fat, less than 10% energy from saturated fatty acids, 55% to 60% energy from carbohydrates, and 15% energy from protein, with a cholesterol intake less than 300 mg/d and fiber intake of 35 g/d or greater.
  Interventions: Dietary Supplement: genistein
- Genistein (Experimental): Genistein 54 mg/day in 2 tablets for 12 months. All participants were counseled on an moderate hypocaloric, Mediterranean-style diet composed of 25% to 30% energy from fat, less than 10% energy from saturated fatty acids, 55% to 60% energy from carbohydrates, and 15% energy from protein, with a cholesterol intake less than 300 mg/d and fiber intake of 35 g/d or greater.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: genistein — pills of 27 mg, twice per day for 12 months
  Arms: Lifestyle counseling
Dietary Supplement: placebo — sugar pills twice per day for 12 months
  Arms: Genistein

SUMMARY:
The purpose of this study is to determine whether the phytoestrogen genistein is effective in improving bone condition in pre-menopausal and post-menopausal women suffering for osteopenia. Since, during the study the investigators realized that at least 70% of post-menopausal recruited women suffered for metabolic syndrome (MS), we have added only in these women, as secondary outcome measures, the evaluation of markers of cardiovascular risk.

DETAILED DESCRIPTION:
MS prevalence increases after the onset of menopause, because of estrogen deficiency. It is still not clear if menopause itself increases the risk of cardiovascular diseases in al women or only in those that develop MS. Many MS patients that show slight modification in cardiovascular and metabolic parameters are not generally pharmacologically treated since diabetes or alteration in the lipid profile are not evidenced. In this respect it is of importance to develop new therapeutic strategies to prevent and treat MS. Genistein (4,5,7-trihydroxyisoflavone), shown a potentially preventive role on the cardiovascular apparatus in post-menopausal women, may be termed as selective ER modulator (SERM), since it reveals both ER-alpha full agonist and ER-beta partial agonist activity.

The investigators studied whether genistein may represent an efficacious and safe alternative for reducing vascular risk in postmenopausal women with metabolic syndrome. The clinical study was a randomized, double-blind, placebo-controlled study involving 150 patients with metabolic syndrome. After a 4-week stabilization on a standard fat-reduced diet, participants were randomly assigned to receive either phytoestrogen genistein (54 mg/day) or placebo for 6 months. At baseline and following treatment fasting plasma glucose, insulin, insulin resistance (HOMA-IR), lipid concentrations, plasma total homocysteine, leptin, adiponectin and visfatin were measured. Bioimpedentiometric and nutritional analysis, as well as a safety assessment of the endometrium and vagina were also performed.

ELIGIBILITY:
Inclusion Criteria:

Post-menopausal satus

The presence of three or more of the five following criteria:

waist circumference ≥88 cm; Triglycerides ≥150 mg/dl or on drug treatment for elevated triglycerides; high-density-lipoprotein (HDL) cholesterol <50 mg/dl or on drug treatment for reduced HDL-C; Fasting glucose ≥100 mg/dl or on drug treatment for elevated glucose; Blood pressure ≥130/85 mmHg or on antihypertensive drug treatment in a subject with a history of hypertension.

Exclusion Criteria:

clinical or laboratory evidence of confounding systemic diseases (e.g., chronic renal or hepatic failure, chronic inflammatory diseases) cardiovascular disease (CVD) defined as documented myocardial infarction, ischaemic heart disease, coronary heart bypass, coronary angioplasty, cerebral thromboembolism, and peripheral amputations, or by Minnesota codes 1°1-3, 4°1-4, 5°1-3 at a standard ECG performed in the 12 months preceding the study; coagulopathy; use of oral or transdermal estrogen, progestin, androgens, selective estrogen receptor modulators, or other steroids; treatment in the preceding six months with polyunsaturated n-3 fatty acids supplements, non steroidal anti-inflammatory drugs (NSAIDs) or steroids, that would interfere with evaluation of the study medication; smoking habit of more than 2 cigarettes daily.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
markers of bone reabsorption: CTX (C-telopeptide of type I collagen ) and of bone formation: bone ALP (Alkaline phosphatase), plus calcaneus ultrasonography variation values | baseline and six months for markers of bone reabsorption, while baseline and 12 months for evaluation of calcaneus ultrasonography variation values
homeostasis model assessment for insulin resistance (HOMA-IR) | change from baseline at 6 and 12 months
  HOMA-IR was calculated using the following formula: fasting glucose (mg/dl) X fasting insulin (uIU/ml)/22.5.

SECONDARY OUTCOMES:
body mass index | baseline, 6 months and 12 months
  The body mass index (BMI) is calculated by dividing the weight measured in kilograms by the square of the height measured in metres [i.e. BMI = Weight (kg)/ Height (m)]2.
Blood pressure | basal, 6 and 12 months
  Three seated blood pressure measurements were taken on the right arm with a sphygmomanometer after the participant had been resting for at least 5 min. Blood pressure values were based on the average of the second and third measurements.
Metabolic variables | basal, 6 and 12 months
  Fasting glucose and insulin were measured in serum collected after an overnight fast using routine methods. Total cholesterol, High Density Lipoprotein-Cholesterol (HDL-C), and triglycerides were measured by using a routine enzymatic method, and the Low-Density Lipoprotein Cholesterol (LDL-C) level was calculated by using the Friedewald formula: [Total cholesterol (mg/dL) - High Density Lipoprotein-Cholesterol (HDL-C) (mg/dL) - triglycerides (mg/dL)/5].
Inflammatory markers | basal, 6 and 12 months
  Serum visfatin, adiponectin, and homocysteine were measured by using an immunoenzymatic assay was measured by using an immunoenzymatic assay.
Adverse events | basal, 6 and 12 months
  Participants were asked about symptoms at clinic visits every 6 months. Standard clinical evaluations and laboratory analyses, including hematologic, renal, and liver function tests, were done every 6 months. Endometrial thickness was evaluated by using ultrasonography at baseline, 6 months, and 1 year. The endometrial thickness was measured in the sagittal plane from 1 basal layer to the other. If the endometrial thickness was 8 mm or greater or if uterine bleeding occurred, hysteroscopy and endometrial biopsy were performed. All unfavorable and unintended clinical effects were considered adverse effects and were evaluated for severity, duration, seriousness, and relation to the study drug and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, professor, Principal Investigator — University of Messina, Italy; Francesco Squadrito, MD, Principal Investigator — University of Messina
Locations (3):
- Italy (3):
  - University of Magnia Graecia, Catanzaro, Italy
  - University of Palermo, Palermo, Italy
  - Azienda Policlinico Universitario, G. Martino, Messina

REFERENCES:
- [Background] Marini H, Minutoli L, Polito F, Bitto A, Altavilla D, Atteritano M, Gaudio A, Mazzaferro S, Frisina A, Frisina N, Lubrano C, Bonaiuto M, D'Anna R, Cannata ML, Corrado F, Adamo EB, Wilson S, Squadrito F. Effects of the phytoestrogen genistein on bone metabolism in osteopenic postmenopausal women: a randomized trial. Ann Intern Med. 2007 Jun 19;146(12):839-47. doi: 10.7326/0003-4819-146-12-200706190-00005. PMID 17577003
- [Background] D'Anna R, Cannata ML, Atteritano M, Cancellieri F, Corrado F, Baviera G, Triolo O, Antico F, Gaudio A, Frisina N, Bitto A, Polito F, Minutoli L, Altavilla D, Marini H, Squadrito F. Effects of the phytoestrogen genistein on hot flushes, endometrium, and vaginal epithelium in postmenopausal women: a 1-year randomized, double-blind, placebo-controlled study. Menopause. 2007 Jul-Aug;14(4):648-55. doi: 10.1097/01.gme.0000248708.60698.98. PMID 17251874
- [Background] Crisafulli A, Altavilla D, Squadrito G, Romeo A, Adamo EB, Marini R, Inferrera MA, Marini H, Bitto A, D'Anna R, Corrado F, Bartolone S, Frisina N, Squadrito F. Effects of the phytoestrogen genistein on the circulating soluble receptor activator of nuclear factor kappaB ligand-osteoprotegerin system in early postmenopausal women. J Clin Endocrinol Metab. 2004 Jan;89(1):188-92. doi: 10.1210/jc.2003-030891. PMID 14715848
- [Background] Morabito N, Crisafulli A, Vergara C, Gaudio A, Lasco A, Frisina N, D'Anna R, Corrado F, Pizzoleo MA, Cincotta M, Altavilla D, Ientile R, Squadrito F. Effects of genistein and hormone-replacement therapy on bone loss in early postmenopausal women: a randomized double-blind placebo-controlled study. J Bone Miner Res. 2002 Oct;17(10):1904-12. doi: 10.1359/jbmr.2002.17.10.1904. PMID 12369794
- [Derived] Irace C, Marini H, Bitto A, Altavilla D, Polito F, Adamo EB, Arcoraci V, Minutoli L, Di Benedetto A, Di Vieste G, de Gregorio C, Gnasso A, Corrao S, Licata G, Squadrito F. Genistein and endothelial function in postmenopausal women with metabolic syndrome. Eur J Clin Invest. 2013 Oct;43(10):1025-31. doi: 10.1111/eci.12139. Epub 2013 Jul 30. PMID 23899172